CLINICAL TRIAL: NCT05414240
Title: A Randomized, Double-blind Placebo-Controlled Study of Ibudilast for Treating Alcohol Use Disorder
Brief Title: Ibudilast for Treating Alcohol Use Disorder
Acronym: Ibudilast
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Henry Kranzler, Professor of Psychiarty, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 851593
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder (AUD); Alcoholism
Keywords: Ibudilast; alcohol
MeSH Terms: conditions — Alcoholism | interventions — ibudilast; Practice Management, Medical

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-groups design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibudilast (Active Comparator): IBUD at a dosage of 20 mg twice daily for 2 days, with an increase to 50 mg twice daily on day 3. The dosage will remain at 50 mg twice daily through most of the rest of the 6-week treatment period. However, for the last three days of week 6, participants will reduce the dosage gradually to 20 mg twice daily prior to discontinuing it at the end of the treatment period.
  Interventions: Drug: Ibudilast; Behavioral: Medical management
- Inactive placebo (Placebo Comparator): Placebo twice daily for 6-week treatment period. Placebo will match active medication in appearance and size.
  Interventions: Behavioral: Medical management; Drug: Placebo

INTERVENTIONS:
Drug: Ibudilast — IBUD at a dosage of 20 mg twice daily for 2 days, with an increase to 50 mg twice daily on day 3. The dosage will remain at 50 mg twice daily through most of the rest of the 6-week treatment period. However, for the last three days of week 6, participants will reduce the dosage gradually to 20 mg twice daily prior to discontinuing it at the end of the treatment period.
  Other Names: MN-166, previously known as AV411 and the formulation is 10-mg delayed-release Pinatos® capsules
  Arms: Ibudilast
Behavioral: Medical management — All subjects receive 6 weeks of medical management (Pettinati et al. 2004) will support subjects efforts to reduce or stop their drinking.
Drug: Placebo — Placebo twice daily for 6-week treatment period. Placebo will match active medication in appearance and size.
  Other Names: Inactive substance
  Arms: Inactive placebo

SUMMARY:
This is a research study involving 6 weeks of study medication, Ibudilast or a placebo (an inactive substance) and medical management counseling to reduce or stop drinking. Ibudilast is not approved by the U.S. FDA for clinical use in the United States, but it is has been used for many years in Japan for its anti-inflammatory effects. Its use in the treatment of alcohol dependence is experimental. By reducing inflammation, Ibudilast may help some people reduce or stop drinking. We have obtained an Investigational New Drug Application (IND) approval for this study from the FDA. Ibudilast has been used clinically for 20 years in Asia for treating bronchial asthma and, more recently, for post-stroke dizziness and ocular allergies and has been shown to be safe and well tolerated.

DETAILED DESCRIPTION:
Study eligibility is determined at an initial screening visit, which can be completed in a single day or divided over multiple days. Portions of the screening may occur by telephone or video conference. Participants are asked not to drink before this and at all study visits. At all study visits, study staff will check breath alcohol level using a breathalyzer. If the breath alcohol level is greater than 0.02% (which can result from a single standard drink), participants may not be able to complete the visit.

Screening Visit: The screening visit will determine whether the study is a good fit for participants. It take about two hours to complete.

* Participants will be asked to show legal photo ID and undergo a breathalyzer test to ensure that the breath alcohol level is below 0.02% to complete this visit. A reading test wil be given to evaluate participant's ability to understand the consent form and study assessment questionnaires.
* Once the informed consent is complete a study clinician will complete a medical history and perform a physical examination. Study staff will draw approximately 3 tablespoons of blood for standard laboratory tests. Participants will also be asked to provide a urine sample to conduct a urinalysis, drug screen, and a urine pregnancy test (only for for women of childbearing potential--i.e., who have not had a hysterectomy, bilateral removal of the ovaries, or a tubal ligation or is less than two years postmenopausal). We will not include women who are pregnant, breast-feeding.
* Eligible participants will be required to provide the names and contact information of one or two people (trusted friends or family members) who may serve as additional contacts to assist staff with locating participants for safety or other study-related reasons.
* Participants will be asked to complete 4 assessments of about psychological health and alcohol and drug use history.

First Study Drug Visit (Week 1): Staff will contact participants within 2 weeks after completing the screening visit to inform eligibility status and schedule the next study visit.

* This visit will take approximately two hours to complete.
* Participants will be asked to complete a breathalyzer test and study staff will measure weight and vital signs (blood pressure and heart rate).
* Woman of childbearing potential, will be asked to provide a urine sample for a pregnancy test.
* Participants will be asked to complete 7 assessments about psychological health and alcohol and drug use history.
* Staff will instruct participants how to use the interactive voice response (IVR) system via telephone. During the 8 weeks of the study, participants will be asked to call a toll-free phone number each day, between 5:00 and 8:00 p.m. to connect to the system. Access to the system via a touch-tone phone requires a study ID and a password. The system has prompts to answer questions about feelings and use of alcohol on the day of the call and the preceding day. It takes about 5 to 8 minutes to complete the daily interview. The IVR system will provide a reminder if a call has not been completed by 8:15 p.m.
* The first brief counseling session will last about 45 minutes. The study nurse will discuss a treatment goal either to drink less or become completely abstinent. The nurse will also encourage participants to consider ways to reduce or stop drinking, based upon the treatment goal.
* Participants will be assigned to receive the study medication from the study clinician, which will be either ibudilast or placebo (an inactive substance). The decision as to which medication received will be random, like a flip of a coin. The ibudilast or placebo will look the same. Neither participants nor any of the study personnel will know which medication is received. In an emergency, though, the study staff in charge of the study medication can be contacted for that information.
* At each visit, study staff will ask about any side effects or other adverse events.

Biweekly Visits (Weeks 2, 3, and 4): At each biweekly visit:

* The staff will check breath alcohol concentration (Breathalyzer), weight, and vital signs and ask about any side effects or other adverse events that were experienced.
* Participants will asked to complete 6 assessments about psychological health and alcohol and drug use history. These should take about 20 minutes to answer.
* Participants will receive brief counseling from the study clinician, which will last about 20 minutes.
* At week 3, woman of childbearing potential, will have another urine pregnancy test. If the urine permanency test is positive, staff will discontinue the medication and the participant will be referred to an obstetrician for care.
* At each visit the study clinician will collect your study medication bottles with any remaining capsules and dispense another week's supply of study medication.
* Participants will continue to call and complete the toll-free IVR number nightly.

  4. Endpoint Visit (End of Week 6): At this visit:
* The staff will measure breath alcohol concentration (Breathalyzer), weight, and vital signs and asked about any side effects or other adverse events that may have experienced.
* The study staff will ask you to complete 9 assessments about your psychological health and your alcohol and drug use history. These should take about 45 minutes to complete.
* Study staff will draw 1 tablespoonful of blood for lab tests.
* Participants will receive brief counseling from the study clinician, which will last about 20 minutes.

Follow-up Visits (4 weeks after endpoint visit): At the follow-up visit (which will take about one hour), the study staff will:

* Check breath alcohol concentration (Breathalyzer), weight and vital signs.
* Draw 1 tablespoonful of blood for lab tests.
* Participants will be asked to complete 9 assessments about psychological health and alcohol and drug use history.
* Once participants have completed the study, they will have an option to receive a letter to inform them whether they received ibudilast or placebo medication.

Early Termination Visit

• Participants who choose to withdraw from the study before participation is complete will be asked to return to the research center for a visit to allow staff to administer the end-of-study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Physically healthy, based on medical history and physical examination and approval of the study physician
2. Meets current DSM-5 criteria for AUD
3. Average weekly ethanol consumption of >24 standard drinks for men and >18 standard drinks for women, with a weekly average of > 2 HDDs during the month before screening
4. Stated goal to reduce drinking to safe levels or to stop drinking
5. Able to read English at an 6th grade or higher level and no gross cognitive impairment
6. Willingness to nominate an individual who will know the subject's whereabouts to facilitate follow up during the study
7. Women of child-bearing potential (i.e., who have not had a hysterectomy, bilateral oophorectomy, tubal ligation or less than two years postmenopausal) must be non-lactating and practicing a reliable method of birth control and have a negative urine pregnancy test prior to the initiation of treatment. Examples of medically acceptable methods for this protocol include: the birth control pill, intrauterine device, injection of Depo-Provera, Norplant, contraceptive patch, contraceptive ring, double-barrier methods (such as condoms and diaphragm/spermicide), male partner sterilization, abstinence (and agreement to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence), and tubal ligation.
8. Willingness to provide signed, informed consent and commit to completing the procedures in the study

Exclusion Criteria:

1. A current, clinically significant physical disease or abnormality based on medical history, physical examination, or routine laboratory evaluation, including direct bilirubin elevations of >110% or a transaminase elevation >300% of normal
2. Current, serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, panic disorder, borderline or antisocial personality disorder, organic mood or mental disorders, eating disorder, or imminent suicide or violence risk)
3. Current DSM-5 diagnosis of dependence on a drug other than alcohol, marijuana or nicotine
4. Current regular treatment with a psychotropic medication (e.g., benzodiazepines, anticonvulsants), which affect neurotransmitter systems, or a medication to treat alcohol dependence. Stable antidepressant treatment for at least 1 month is acceptable.
5. Urine drug screen positive for recent use of opioids, cocaine, or amphetamines (may be repeated once and if the result is negative on repeat it is not exclusionary)
6. Judged by the principal investigator or his designee to be an unsuitable candidate for receipt of an investigational drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the frequency of heavy drinking | 6-week treatment period.
  Frequency of heavy drinking (defined as 4 or more drinks in a day for women and five or more drinks in a day for men).

SECONDARY OUTCOMES:
Change in the number of abstinent days, heavy drinking days during the last month of treatment. | 6-week treatment period.
  Change in the number of abstinent days, absence of any heavy drinking days during the last month of treatment, mean daily alcohol consumption, drinks/drinking day.

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Kranzler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States